CLINICAL TRIAL: NCT01679522
Title: Prospective Randomized Comparison of Single-port and Four-port Laparoscopic Staging Operation for Endometrial Cancer
Brief Title: Feasibility Study of Laparoendoscopic Single Site Surgical Staging for Endometrial Cancer
Acronym: LESS-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LESS-E
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; laparoscopic surgical staging; single-port; four-port
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-port surgery group (Experimental): Single-port laparoscopic surgical staging including total hysterectomy, pelvic lymph node dissection, and/or bilateral salpingooophorectomy, and/or para-aortic lymph node dissection
  Interventions: Procedure: single-port laparoscopic surgical staging
- Four-port surgery group (Active Comparator): Four-port laparoscopic surgical staging including total hysterectomy, pelvic lymph node dissection, and/or bilateral salpingooophorectomy, and/or para-aortic lymph node dissection
  Interventions: Procedure: Four-port laparoscopic surgical staging

INTERVENTIONS:
Procedure: single-port laparoscopic surgical staging — single-port laparoscopic surgical staging indluding total hysterectomy, pelvic lymph node dissection, and/or bilateral salpingooophorectomy, and/or para-aortic lymph node dissection
  Arms: Single-port surgery group
Procedure: Four-port laparoscopic surgical staging — Four-port laparoscopic surgical staging indluding total hysterectomy, pelvic lymph node dissection, and/or bilateral salpingooophorectomy, and/or para-aortic lymph node dissection
  Arms: Four-port surgery group

SUMMARY:
To compare the feasibility, safety, and efficacy between single-port and four-port laparoscopic surgical staging in patients with early stage endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed endometrial cancer
* Presumed FIGO stage 1
* Endometrioid adenocarcinoma
* patient who is planned to undergo surgical staging
* adequate oran function

  1. WBC > 3000 cells/mcl
  2. Platelets > 100000/mcl
  3. Creatinine < 2.0 mg/dL
  4. Bilirubin < 1.5 * normal and SGOT or SGPT < 3 * normal
* American Society of Anesthesiologists Physical Status I-II
* Eastern Cooperative Oncology Group performance status 0-2
* Patients who have signed an approved Informed Consent

Exclusion Criteria:

* Uncontrolled medical disease
* Active infectious disease requiring antibiotics
* Previous pelvic radiation therapy
* Pregnant and lactating woman
* Patient who requires additional surgical procedures which are not necessary for surgical staging of endometrial cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
operating time | 1 day (Immediately after operation)
  Total operation time and time required for each procedure are calculated and compared.
Number of lymph nodes retrieved | 1 week after surgery
  The number of right pelvic lymph nodes and left pelvic lymph nodes were obtained and compared.

SECONDARY OUTCOMES:
Postoperative pain | within 1 week after surgery
  The VAS pain score was obtained every 8 hours after surgery and compared.
Postoperative analgesics requirement | within 1 week after surgery
  If the VAS pain score is 3 or more or the patient desires, additional pain medication is administered. The frequency of the pain medication administered in this way is investigated and compared.
transfusion requirement and amount | within 1 week after surgery
  Investigate and compare blood transfusion volume and frequency during and after surgery.
postoperative complications | within 1 month after surgery
  Compare the frequency of fever, urinary retention, anemia, and nausea after surgery.
recurrence free survival | 34 months after surgery
  Compare RFS during the follow-up period.
overall survival | 34 months after surgery
  Compare OS during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang OJ, Nam JH, Park JY. Laparo-endoscopic single-site versus conventional laparoscopic surgery for early-stage endometrial cancer: A randomized controlled non-inferiority trial. Gynecol Oncol. 2023 Jun;173:74-80. doi: 10.1016/j.ygyno.2023.04.005. Epub 2023 Apr 25. PMID 37105060